CLINICAL TRIAL: NCT02425852
Title: A Randomized, Multicenter Open Label Study Comparing Early Administration of Azathioprine Plus Infliximab to Corticosteroids Plus Azathioprine for Acute Severe Colitis
Brief Title: A Randomized, Multicenter Open Label Study Comparing Early Administration of Azathioprine Plus IFX to Steroids Plus Azathioprine for Acute Severe Colitis
Acronym: ACTIVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GETAID 2015-02
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Azathioprine; Infliximab; Prednisolone; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination therapy arm (Active Comparator): Infliximab 5 mg/kg plus Azathioprine 2-2.5 mg/kg/day. Azathioprine will be introduced at day 5-7 and continued until week 52. Azathioprine dose regimen will be between 2 and 2.5 mg/kg/d, as close as possible to 2.5 mg/kg/d, or to 1.5 mg/kg/d for 6-mercaptopurine, in one daily intake.
  Interventions: Drug: Azathioprine; Drug: Infliximab
- Azathioprine arm (Active Comparator): Intravenous steroids will be continue until day 2. Then, steroid therapy will be orally administered at a dose of 40-60 mg/day ou 1 mg/kg/day prednisolone (or equivalent) and progressively reduced by 10mg step every week to 20mg per day, and then reduced by 5mg step every week until stopped. Hydrocortisone intake to prevent steroid weaning will be authorized until supradrenal function normalization.
  In patients with clinical response at day 7, Azathioprine will be introduced at day 5-7 and continued until week 52. Azathioprine dose regimen will be between 2 and 2.5 mg/kg/d, as close as possible of 2.5 mg/kg/d, or of 1.5 mg/kg/d for 6-mercaptopurine, in one daily intake.
  Interventions: Drug: Azathioprine; Drug: Prednisolone; Drug: Hydrocortisone

INTERVENTIONS:
Drug: Azathioprine — Azathioprine alone versus Azathioprine and IFX
Drug: Infliximab
  Arms: Combination therapy arm
Drug: Prednisolone
  Arms: Azathioprine arm
Drug: Hydrocortisone
  Arms: Azathioprine arm

SUMMARY:
PHASE : IV TYPE OF STUDY : With direct benefit. DESCRIPTIVE : Multicentre, randomized, open label study. INCLUSION CRITERIA : Acute severe ulcerative colitis. OBJECTIVES : To compare the efficacy and safety of early administration of the combination therapy with infliximab and azathioprine with steroids and azathioprine in patients with acute severe ulcerative colitis treated with intravenous steroids.

STUDY TREATMENTS : All patients :

Intravenous steroids (0.8 mg/kg/day of methylprednisolone or equivalent) for 5 days.

Combination therapy arm:

Infliximab 5 mg/kg plus Azathioprine 2-2.5 mg/kg/day.

Azathioprine arm:

Steroids tapering for 3 months and Azathioprine 2-2.5 mg/kg/day.

DETAILED DESCRIPTION:
NUMBER OF PATIENTS : 73 patients in each group i.e. a total of 146patients. RECRUITMENT PERIOD : 36 months STUDY DURATION : 12 months

PRIMARY END POINT : Treatment failure is defined by:

* Absence of steroid-free remission at W52 according to the total Mayo Disease Activity Index score
* OR Absence of mucosal healing (Mayo endoscopic subscore 0-1)
* OR Adverse event leading to treatment interruption
* OR Colectomy
* OR Death
* OR Infliximab withdrawal in the combination therapy group OR Infliximab introduction in the azathioprine group SECONDARY END POINT: - Clinical response and remission at D7, W14 and W52 (according to Lichtiger score and total Mayo Disease Activity Index score)
* Endoscopic and histological response
* Mucosal healing (partial endoscopic Mayo subscore 0)
* Colectomy rate
* Adverse events rate
* Fecal calprotectin
* Health-economic outcome

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Diagnosis of UC according to Lennard-Jones criteria (Appendix 1).
* Endoscopically demonstrated colorectal lesions localized above the anal margin and extending at least up to 15cm proximally (Endoscopic Mayo subscore ≥ 2).
* Acute flare requiring hospitalization
* Severe acute flare of UC with a Lichtiger Index score > 10 at Day -3
* Adequate contraception for male or female subjects of childbearing potential, which will be continued throughout the study and at least 3 months after study termination.

3.2 EXCLUSION CRITERIA

* Pregnant or breast-feeding woman.
* Previous treatment with infliximab.
* Treatment with adalimumab or golimumab within 8 weeks before randomization
* Treatment with vedolizumab within 4 weeks before randomization
* Azathioprine or 6-mercaptopurine treatment initiated more than 4 weeks before screening.
* Ongoing intravenous steroids for more than 96 hours at time of the screening
* Contraindication for anti-TNF therapy
* Indication for immediate surgery.
* History of colorectal dysplasia.
* Diagnosis of Crohn's disease or indeterminate colitis
* Positive stool tests for amoebiasis and/or positive bacteriological culture for Salmonella, Shigella, Yersinia and Campylobacter and/or presence of Clostridium difficile B toxin in the stools.
* Renal failure (creatininemia > upper limit of normal laboratory value).
* Uncontrolled high blood pressure.
* HIV, HBV viral infection (except the presence of positive anti-HBs antibodies) with serology not older than 3 months.
* Uncontrolled bacterial or active viral infection.
* Past medical history of malignant condition in the last 5 years (including leukaemia, lymphoma and myelodysplasia) except for baso-cellular cutaneous cancers.
* Past medical history of myocardial infarction or heart failure.
* Intradermal reaction to Tuberculin (Tubertest® 5 units) > 5mm or positive interferon-gamma release assay (Quantiferon®)
* Active tuberculosis
* Untreated latent tuberculosis (see national recommendations. Appendix 2).
* Abnormal blood count with polynuclear neutrophils < 1,500 G/L or white cells < 3,000, or platelets < 100,000 G/L.
* Unexplained rise higher than 3 times the normal level for transaminases, alkaline phosphatases and/or higher than twice the normal level for bilirubin.
* Severe acute or chronic medical or psychiatric condition that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in judgement of the investigator, would make the subject inappropriate for entry in this study.
* Subjects who, in the opinion of the investigator, will be uncooperative or unable to comply with study procedures.
* Participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with treatment failure at week 52. | Week 52
  Failure is defined as:
  * absence of steroid-free remission (Total Mayo Disease Activity Index (DAI) score ≤ 2 with no individual subscore > 1)
  * absence of mucosal healing (Endoscopic Mayo DAI subscore ≤ 1)
  * or severe adverse event leading to treatment interruption between day 0 and week 52
  * or colectomy between day 0 and week 52
  * or fatality between day 0 and week 52
  * or infliximab withdrawal for failure and /or intolerance in the combination therapy group
  * or any biological agent introduction in the azathioprine group

SECONDARY OUTCOMES:
Percentage of patients in clinical response at day 7 | 7 days
  Percentage of patients in clinical response at day 7 (Lichtiger Index score<10 with a decrease of at least 3 points compared with the baseline score) and at week 14 and week 52 (a decrease from baseline in the Mayo score ≥30% and ≥3 points, accompanied by either a rectal bleeding subscore of 0 or 1 or a decrease from baseline in the rectal bleeding subscore ≥1)
  - Percentage of patients in clinical remission at day 7, week 14 and week 52

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien Amiot, MD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives; Laurent Peyrin-Biroulet, MD, PhD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives
Locations (16):
- France (16):
  - Chu Besancon, Besançon
  - CHU de CLERMONT FERRAND- Hopital Estain, Clermont-Ferrand
  - APHP- Hopital BEAUJON, Clichy
  - Hopital Louis Mourrier, Colombes
  - Henri Mondor Hospital, Créteil
  - Chu Kremlin Bicetre, Le Kremlin-Bicêtre
  - CHRU Lille, Lille
  - Chu Montpellier, Montpellier
  - CHU de NICE- Hopital Archet 2, Nice
  - Hopital Saint Louis, Paris
  - Hopital St Antoine, Paris
  - Hopital Saint Joseph, Paris
  - CHU RENNES - Hopital Pontchaillou, Rennes
  - Chu Rouen, Rouen
  - Chu Saint Etienne, Saint-Etienne
  - CHU NANCY - Hopital Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Amiot A, Seksik P, Meyer A, Stefanescu C, Wils P, Altwegg R, Vuitton L, Plastaras L, Nicolau A, Pereira B, Duveau N, Laharie D, Mboup B, Boualit M, Allez M, Rajca S, Chanteloup E, Bouguen G, Bazin T, Goutorbe F, Richard N, Moussata D, Vicaut E, Peyrin-Biroulet L. Top-down infliximab plus azathioprine versus azathioprine alone in patients with acute severe ulcerative colitis responsive to intravenous steroids: a parallel, open-label randomised controlled trial, the ACTIVE trial. Gut. 2025 Jan 17;74(2):197-205. doi: 10.1136/gutjnl-2024-333281. PMID 39586616